CLINICAL TRIAL: NCT00203658
Title: LITE Study, Appendix A (HOME-LITE), Amendment 6
Brief Title: Assessment of Long-Term Out-of-Hospital Treatment of Patients With Proximal Deep Vein Thrombosis (DVT) Using Low-Molecular-Weight Heparin (LMWH) Versus LMWH Followed by Warfarin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); LEO Pharma (Industry); Dupont Applied Biosciences (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 2736-2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2005-09

CONDITIONS: Thrombosis; Thromboembolism; Venous Thrombosis
MeSH Terms: conditions — Thrombosis; Thromboembolism; Venous Thrombosis | interventions — Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin sodium

SUMMARY:
The purpose of this study is to assess the long-term out-of-hospital treatment of patients with proximal venous thrombosis through the administration of subcutaneous low-molecular-weight heparin (tinzaparin sodium) versus low-molecular-weight heparin followed by warfarin sodium.

DETAILED DESCRIPTION:
Two studies demonstrated that out-of-hospital low-molecular-weight heparin given by twice daily subcutaneous injection without laboratory monitoring was as effective and as safe as continuous intravenous heparin given in-hospital. Innohep (tinzaparin) has been shown to be safe and effective for both the initial and long-term treatment of DVT. The Home LITE study compares long-term Innohep treatment to treatment with a combination of initial low-molecular-weight heparin followed by standard long-term warfarin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a first or recurrent episode of acute proximal vein thrombosis who are eligible for outpatient or home care during the initial therapy.

Exclusion Criteria:

* Any condition which, in the opinion of the investigator, precludes entire out-of-hospital treatment
* Presence of familial bleeding diathesis or the presence of active bleeding contraindicating anticoagulant therapy
* Receiving therapeutic heparin for more than 48 hours or have already been on warfarin for more than 2 days for the treatment of proximal deep vein thrombosis
* Receiving long-term warfarin treatment
* Females who are pregnant
* Known allergy to heparin, warfarin sodium, or bisulfites
* History of heparin-associated thrombocytopenia
* Severe malignant hypertension
* Hepatic encephalopathy
* Severe renal failure
* Inability to attend follow-up due to geographic inaccessibility
* Inability or refusal to give signed informed consent
* Mothers who are breast-feeding and who are unable to refuse to discontinue breast-feeding during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1997-04; Study Completion 2000-10

PRIMARY OUTCOMES:
objectively documented recurrent venous thromboembolism during initial treatment or during the 12 week follow-up period
death during initial treatment or during the 12 week follow-up period
safety endpoint for assessing harm was the occurrence of bleeding (all, major or minor) during the 12 week treatment interval

SECONDARY OUTCOMES:
recurrent venous thromboembolism at 12 months
death at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell D Hull, MBBS, MSc, Principal Investigator — University of Calgary
Locations (1):
- Thrombosis Research Unit, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Koopman MM, Prandoni P, Piovella F, Ockelford PA, Brandjes DP, van der Meer J, Gallus AS, Simonneau G, Chesterman CH, Prins MH. Treatment of venous thrombosis with intravenous unfractionated heparin administered in the hospital as compared with subcutaneous low-molecular-weight heparin administered at home. The Tasman Study Group. N Engl J Med. 1996 Mar 14;334(11):682-7. doi: 10.1056/NEJM199603143341102. PMID 8594426
- [Background] Levine M, Gent M, Hirsh J, Leclerc J, Anderson D, Weitz J, Ginsberg J, Turpie AG, Demers C, Kovacs M. A comparison of low-molecular-weight heparin administered primarily at home with unfractionated heparin administered in the hospital for proximal deep-vein thrombosis. N Engl J Med. 1996 Mar 14;334(11):677-81. doi: 10.1056/NEJM199603143341101. PMID 8594425
- [Background] Lancaster TR, Singer DE, Sheehan MA, Oertel LB, Maraventano SW, Hughes RA, Kistler JP. The impact of long-term warfarin therapy on quality of life. Evidence from a randomized trial. Boston Area Anticoagulation Trial for Atrial Fibrillation Investigators. Arch Intern Med. 1991 Oct;151(10):1944-9. PMID 1929681
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798